CLINICAL TRIAL: NCT06321562
Title: A First-In-Human, Open-Label, Dose Escalating, Non-Randomized Study to Assess the Safety and Tolerability of a New Timolol Sustained Release Intraocular Implant (TimoD) in Subjects With Primary Open Angle Glaucoma With Pseudophakia
Brief Title: Safety and Tolerability of a Timolol Releasing Intraocular Implant in Subjects With Primary Open-angle Glaucoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to the difficulties to enrol participant
Sponsor: EyeD Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: EyeD-010-003; 2024-511254-51-00 (EU CTIS Number); CIV-21-12-038426 (Other: EUDAMED)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Glaucoma; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: TimoD implant-Dose 1 (low dose) (Experimental): Participants in the Group 1 will receive a low dose of TimoD implant in the study eye on Day 1.
  Interventions: Drug: TimoD implant; Device: Injector system
- Group 2: TimoD implant-Dose 2 (intermediate dose) (Experimental): Participants in Group 2 will receive an intermediate dose of TimoD implant in the study eye on Day 1 if all participants in Group 1 have completed a 4-week treatment period with the lowest dose of TimoD implant, providing there are no safety issues in Group 1.
  Interventions: Drug: TimoD implant; Device: Injector system
- Group3: TimoD implant-Dose 3 (high dose) (Experimental): Participants in Group 3 will receive a high dose of TimoD implant in the study eye on Day 1 if all participants in Group 2 have completed a 4-week treatment period with the intermediate dose, providing there are no safety issues in Group 2.
  Interventions: Drug: TimoD implant; Device: Injector system

INTERVENTIONS:
Drug: TimoD implant — Consists of 1 TimoD implant administration in the study eye
  Other Names: Intraocular implant releasing timolol; Investigational drug
Device: Injector system — This is a CE-marked injector intended for intraocular lens (IOL) delivery. In this study, the injector is used as an"intraocular implant injection system" outside of its scope of intended use.
  Other Names: ACCUJECT™ 2.2.-BL; Investigational device

SUMMARY:
The purpose of this study is to test a new method to deliver an approved medicine called Timolol in the eye of participants with glaucoma and pseudophakia (currently present or to be performed during the concomitant implantation surgery in subjects with age-related cataract eligible to intra-capsular IOL placement). The main questions it aims to answer are how safe the investigational drug is and how the body tolerates it.

The study will also check:

* how safely the implant is placed in and removed from the eye and how the body responds to the procedure,
* how safe different doses of timolol are and how the body handles taking it,
* the amount of Timolol released in the bloodstream,
* if there is any positive effect on the pressure inside the eye.

DETAILED DESCRIPTION:
Timolol will be delivered through an investigational drug called 'TimoD implant'. This implant is placed inside one eye, the study eye, with the help of an instrument (investigational device) called an injector system.

Three dose ranges of TimoD implant will be tested (low, intermediate, and high) in 3 groups of 6 participants.

The Timolol will be released slowly through the implant for up to 1 year (main phase).

Approximately 1 year after the TimoD implant is placed into the eye and in absence of contraindications, the participants will be invited to continue the study in an extension phase. If the participants agree to enter the extension phase and the study investigator confirms it is safe for them, the TimoD implant will remain in the study eye for one additional year.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* In good general and mental health without ongoing clinically significant abnormalities in medical history.
* Clinically proven diagnosis of primary open-angle glaucoma (POAG) in the previous 12 months.
* Subjects with IOP not adequately controlled with the standard medication.
* Pseudophakia.

Exclusion Criteria:

* Concomitant treatment with timolol (systemic), corticosteroids, cytochrome P450 2D6 inhibitors, or α2-agonists.
* Subjects with a history of hypersensitivity or contraindications to β-blockers.
* Significant risks caused by washout of ocular hypotensive medications.
* History of any glaucoma not specified as POAG.
* History of elevated IOP due to corticosteroid use.
* History of ocular trauma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Number and proportion of participants experiencing one or more serious adverse events (SAEs) | From screening visit (up to Day -41) to end of study (Week 108)
Number and proportion of participants experiencing one or more treatment-emergent adverse events (TEAEs) overall and by dose group | From screening visit (up to Day -41) to end of study (Week 108)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Breyer, Kaymak & Klabe Augenchirurgie, Düsseldorf
  - Universitäts-Augenklinik Heidelberg, Heidelberg
  - Universitätsaugenklinik Magdeburg, Magdeburg
  - Augenklinik Sulzbach, Sulzbach
  - Universitäts-Augenklinik Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No